CLINICAL TRIAL: NCT02329860
Title: A Randomized, Double Blind, Placebo Controlled, Multicenter Phase III Study (AHELP) of Apatinib in Patients With Hepatocellular Carcinoma After Systemic Therapy（Chemotherapy and/or Targeted Therapy）
Brief Title: Study of Apatinib After Systemic Therapy in Patients With Hepatocellular Carcinoma(AHELP)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Collaborators: NanJing PLA 81 Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: APTN-III-HCC
Record Dates: First submitted 2014-12-30; First posted 2015-01-01 (Estimated); Results first posted 2024-01-22 (Actual); Last update posted 2024-01-22 (Actual); Status verified 2017-07

CONDITIONS: Carcinoma, Hepatocellular
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — apatinib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Apatinib (Experimental): 750 mg orally (p.o.) every day (qd), 28 days as one cycle
  Interventions: Drug: Apatinib
- Placebo (Placebo Comparator): orally (p.o.) every day (qd), 28 days as one cycle
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Apatinib
  Arms: Apatinib
Drug: Placebo
  Arms: Placebo

SUMMARY:
This was a multicenter, randomized, double-blind, phase III trial. This clinical study evaluates the efficacy and safety of Apatinib in patients with advanced liver cancer who have progressed on Systemic Therapy (Chemotherapy and/or Targeted Therapy).

Approximately 400 patients who meet the entry criteria will be randomly assigned in a 2:1 ratio to Apatinib or placebo (1/3 chance to receive placebo).

Primary endpoint of the study is overall survival.

ELIGIBILITY:
Inclusion Criteria:

1. ≥ 18 years old.
2. Conform to the clinical diagnosis standard strictly or histological or cytological confirmation of HCC (hepatocellular carcinoma) who cannot benefit from treatments of established efficacy with higher priority such as resection, local ablation,and with at least one uni-dimensional measurable lesion by computed tomography (CT) scan or magnetic resonance imaging (MRI) according to RECIST 1.1.
3. Failure or intolerance to prior treatment with chemotherapy and/or targeted therapy (Failure is defined as documented radiological progression according to the radiology charter. Intolerance is defined as ≥ grade 4 hematologic toxicities, ≥ grade 3 non-hematologic toxicities ≥ grade 2 heart, liver or kidney damage).
4. Systemic therapy must have been completed ≥2 weeks before randomization (AEs due to prior treatment ≤ grade 1).
5. Liver function status Child-Pugh Class A or B (score≤7).
6. Barcelona Clinic Liver Cancer stage Category B or C.
7. Eastern Cooperative Oncology Group Performance Status of 0 or 1 within 1 week before randomization.
8. Life expectancy of at least 12 weeks.
9. HBV DNA ≤ 2000IU/ml or 1×10E+4 copy/ml.
10. Adequate bone marrow, liver and renal function as assessed by the following laboratory tests conducted within 1 week before randomization.

    HB ≥ 90g/L; ANC≥1.5×10E+9/L; PLT≥80×10E+9/L; ALB ≥ 29g/L; ALT and AST < 5×ULN; TBIL ≤1.5×ULN; Cr ≤1.5×ULN
11. Women of childbearing potential and men must agree to use adequate contraception .

Exclusion Criteria:

1. Any local treatment (included but not limited: resection, radiotherapy, TAE, TACE, TAI, RFA or PEI) within 4 weeks of randomization.
2. Known hepatic duct carcinoma, mixed cell carcinoma or fibrolamellar hepatocellular carcinoma, known history or suffering from other cancer(except of cured skin basal cell carcinoma or carcinoma in situ of cervix).
3. Patients who will receive liver transplantation.
4. Ascites with clinical symptoms, i.e. require Abdominal paracentesis or drainage treatment such as or Child-Pugh Score>2.
5. Hypertension and unable to be controlled within normal level following treatment of anti-hypertension agents (systolic blood pressure > 140 mmHg, diastolic blood pressure > 90 mmHg).
6. Suffered from grade II or above myocardial ischemia or myocardial infarction, uncontrolled arrhythmias (including QT interval male ≥ 450 ms, female≥ 470 ms).
7. Grade III-IV cardiac insufficiency, according to NYHA criteria or echocardiography check: LVEF<50%.
8. Factors to affect oral administration（such as Patients unable to swallow oral medications, chronic diarrhea and ileus etc. situations evidently affect drug oral medication and absorption）.
9. Previous digestive tract bleeding history within 6 months or evident gastrointestinal bleeding tendency, such as,：Esophageal varices with bleeding risk, local active ulcerative lesions, fecal occult blood≥（++）；if fecal occult blood（+），gastroscope check is required.
10. The Within 28 days ahead of randomization, experience abdomen fistula, gastrointestinal perforation, or abdominal abscess
11. Coagulation abnormalities (INR > 1.5 x ULN, or PT > ULN +4 seconds), with bleeding tendency or are receiving thrombolytic or anticoagulant therapy;
12. Occurrence of central nervous system metastatic or known brain metastatic;
13. Objective evidence of previous or current pulmonary fibrosis history, interstitial pneumonia, Pneumoconiosis, radiation pneumonitis, drug-related pneumonia, Pulmonary function damaged seriously etc.
14. Proteinuria ≥ (++) or 24 hours total urine protein > 1.0 g.
15. Received powerful inhibitor of CYP3A4 within 7 days or powerful inducer of CYP3A4 within 12 days before randomization.
16. Pregnant or breast-feeding women; patients with fertility will not or there is no way to adopt effective contraceptive measures.
17. Mental disorders history, or Psychotropic drug abuse history.
18. Patients who has bone metastasis, has received Palliative radiotherapy (radiotherapy area > 5% marrow area).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Actual)
Dates: Start 2014-03-26 (Actual); Primary Completion 2017-12-15 (Actual); Study Completion 2019-08-14 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Jiangsu hengrui medicine CO. LTD, Lianyungang, Jiangsu, China

REFERENCES:
- [Derived] Qin S, Li Q, Gu S, Chen X, Lin L, Wang Z, Xu A, Chen X, Zhou C, Ren Z, Yang L, Xu L, Bai Y, Chen L, Li J, Pan H, Cao B, Fang W, Wu W, Wang G, Cheng Y, Yu Z, Zhu X, Jiang D, Lu Y, Wang H, Xu J, Bai L, Liu Y, Lin H, Wu C, Zhang Y, Yan P, Jin C, Zou J. Apatinib as second-line or later therapy in patients with advanced hepatocellular carcinoma (AHELP): a multicentre, double-blind, randomised, placebo-controlled, phase 3 trial. Lancet Gastroenterol Hepatol. 2021 Jul;6(7):559-568. doi: 10.1016/S2468-1253(21)00109-6. Epub 2021 May 8. PMID 33971141

RESULTS

PARTICIPANT FLOW:
Groups:
- Apatinib: 750 mg orally (p.o.) every day (qd), 28 days as one cycle
  Apatinib
- Placebo: orally (p.o.) every day (qd), 28 days as one cycle
  Placebo
Period: Overall Study
Arm/Group | Apatinib | Placebo
Started | 267 | 133
Treated | 261 | 132
Completed | 161 | 107
Not Completed | 106 | 26

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Apatinib | Placebo | Total
Number analyzed (Participants) | 261 | 132 | 393
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.8 (10.7) | 50.3 (10.9) | 50.7 (10.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 38 | 16 | 54
  Male | 223 | 116 | 339
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 261 | 132 | 393
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  China | 261 | 132 | 393

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival
Time Frame: Approximately 36 months
Population: The primary efficacy endpoint was analyzed in FAS.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Apatinib | Placebo
Number analyzed (Participants) | 261 | 132
months | 8.7 [7.5 to 9.8] | 6.8 [5.7 to 9.1]

2. Secondary Outcome: Time to Progression（TTP）
Time Frame: Approximately 36 months
Population: The secondary efficacy endpoint was analyzed in FAS.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Apatinib | Placebo
Number analyzed (Participants) | 261 | 132
months | 4.7 [4.5 to 4.8] | 1.9 [1.9 to 2.0]

3. Secondary Outcome: Progression Free Survival (PFS)
Time Frame: Approximately 36 months
Population: [The secondary efficacy endpoint was analyzed in FAS.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Apatinib | Placebo
Number analyzed (Participants) | 261 | 132
months | 4.5 [3.9 to 4.7] | 1.9 [1.9 to 2.0]

4. Secondary Outcome: Objective Response Rate
Time Frame: Approximately 36 months
Population: The secondary efficacy endpoint was analyzed in FAS
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Apatinib | Placebo
Number analyzed (Participants) | 261 | 132
percentage of participants | 10.7 [7.2 to 15.1] | 1.5 [0.2 to 5.4]

5. Secondary Outcome: Disease Control Rate
Time Frame: Approximately 36 months
Population: The secondary efficacy endpoint was analyzed in FAS.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Apatinib | Placebo
Number analyzed (Participants) | 261 | 132
percentage of participants | 61.3 [55.1 to 67.2] | 28.8 [21.2 to 37.3]

ADVERSE EVENTS:
Time Frame: approximately 5 years
Description: Same event may appear as both an adverse event (AE) and serious adverse event (SAE). However, what is presented are distinct events. An event may be categorized as serious in one participant and as non-serious in another, or a participant may have experienced both a serious and non-serious event.
Arm/Group | Apatinib | Placebo
All-Cause Mortality (participants affected / at risk) | 24/257 | 13/130
Serious Adverse Events (participants affected / at risk) | 95/257 | 30/130
Other Adverse Events (participants affected / at risk) | 251/257 | 110/130
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Apatinib (N=257) | Placebo (N=130)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 13 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 5 | 0
Diarrhoea (Gastrointestinal disorders) | 3 | 1
Abdominal pain upper (Gastrointestinal disorders) | 2 | 0
Melaena (Gastrointestinal disorders) | 1 | 1
Vomiting (Gastrointestinal disorders) | 2 | 0
Abdominal distension (Gastrointestinal disorders) | 1 | 0
Duodenal ulcer (Gastrointestinal disorders) | 1 | 0
Gastritis (Gastrointestinal disorders) | 1 | 0
Intestinal obstruction (Gastrointestinal disorders) | 1 | 0
Mouth ulceration (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 0
Death (General disorders) | 8 | 9
Multiple organ dysfunction syndrome (General disorders) | 3 | 1
Pyrexia (General disorders) | 2 | 2
Fatigue (General disorders) | 2 | 0
Asthenia (General disorders) | 1 | 0
Disease progression (General disorders) | 1 | 0
Hepatic encephalopathy (Nervous system disorders) | 7 | 1
Cerebral haemorrhage (Nervous system disorders) | 2 | 0
Encephalopathy (Nervous system disorders) | 2 | 0
Headache (Nervous system disorders) | 2 | 0
Brain stem haemorrhage (Nervous system disorders) | 1 | 0
Dizziness (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 1 | 0
Lung infection (Infections and infestations) | 8 | 1
Gastroenteritis (Infections and infestations) | 2 | 0
Biliary tract infection (Infections and infestations) | 1 | 0
Gingivitis (Infections and infestations) | 1 | 0
Peritonitis (Infections and infestations) | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 0
Hepatic function abnormal (Hepatobiliary disorders) | 4 | 1
Hepatic failure (Hepatobiliary disorders) | 1 | 2
Cholecystitis (Hepatobiliary disorders) | 2 | 0
Perihepatic discomfort (Hepatobiliary disorders) | 1 | 1
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 4 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Bronchial haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Overdose (Injury, poisoning and procedural complications) | 7 | 2
Fibula fracture (Injury, poisoning and procedural complications) | 0 | 1
Post procedural bile leak (Injury, poisoning and procedural complications) | 0 | 1
Toxicity to various agents (Injury, poisoning and procedural complications) | 0 | 1
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Tumour rupture (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Haematuria (Renal and urinary disorders) | 4 | 0
Proteinuria (Renal and urinary disorders) | 3 | 0
Renal hydrocele (Renal and urinary disorders) | 1 | 0
Aspartate aminotransferase increased (Investigations) | 3 | 0
Blood bilirubin increased (Investigations) | 1 | 1
Bilirubin conjugated increased (Investigations) | 0 | 1
Blood phosphorus decreased (Investigations) | 1 | 0
Blood sodium decreased (Investigations) | 1 | 0
Platelet count decreased (Investigations) | 1 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 2 | 0
Electrolyte imbalance (Metabolism and nutrition disorders) | 1 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0
Anaemia (Blood and lymphatic system disorders) | 1 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 0
Acute coronary syndrome (Cardiac disorders) | 0 | 1
Palpitations (Cardiac disorders) | 1 | 0
Sinus bradycardia (Cardiac disorders) | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Hypertension (Vascular disorders) | 2 | 0
Secondary hypertension (Vascular disorders) | 1 | 0
Acquired hydrocele (Reproductive system and breast disorders) | 1 | 0
Vaginal haemorrhage (Reproductive system and breast disorders) | 1 | 0
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Apatinib (N=257) | Placebo (N=130)
Anaemia (Blood and lymphatic system disorders) | 30 | 13
Diarrhoea (Gastrointestinal disorders) | 105 | 21
Vomiting (Gastrointestinal disorders) | 70 | 16
Nausea (Gastrointestinal disorders) | 60 | 12
Abdominal pain (Gastrointestinal disorders) | 54 | 16
Abdominal pain upper (Gastrointestinal disorders) | 49 | 12
Abdominal distension (Gastrointestinal disorders) | 48 | 19
Mouth ulceration (Gastrointestinal disorders) | 28 | 1
Constipation (Gastrointestinal disorders) | 26 | 4
Stomatitis (Gastrointestinal disorders) | 19 | 3
Gingival pain (Gastrointestinal disorders) | 13 | 1
Asthenia (General disorders) | 85 | 23
Pyrexia (General disorders) | 42 | 9
Oedema peripheral (General disorders) | 23 | 9
Fatigue (General disorders) | 22 | 4
Chest pain (General disorders) | 19 | 2
Upper respiratory tract infection (Infections and infestations) | 23 | 8
Platelet count decreased (Investigations) | 143 | 23
Aspartate aminotransferase increased (Investigations) | 136 | 43
Blood bilirubin increased (Investigations) | 133 | 40
White blood cell count decreased (Investigations) | 105 | 10
Neutrophil count decreased (Investigations) | 97 | 10
Alanine aminotransferase increased (Investigations) | 88 | 28
Bilirubin conjugated increased (Investigations) | 83 | 18
Gamma-glutamyltransferase increased (Investigations) | 53 | 25
Protein urine present (Investigations) | 53 | 8
Blood bilirubin unconjugated increased (Investigations) | 40 | 6
Blood pressure increased (Investigations) | 39 | 5
Blood lactate dehydrogenase increased (Investigations) | 33 | 9
Blood alkaline phosphatase increased (Investigations) | 30 | 13
Blood urine present (Investigations) | 27 | 6
Haemoglobin decreased (Investigations) | 21 | 2
Weight decreased (Investigations) | 21 | 6
Urobilinogen urine increased (Investigations) | 20 | 7
Blood albumin decreased (Investigations) | 19 | 4
Red blood cells urine positive (Investigations) | 19 | 5
White blood cells urine positive (Investigations) | 16 | 5
Urine bilirubin increased (Investigations) | 14 | 4
Protein total decreased (Investigations) | 13 | 3
Decreased appetite (Metabolism and nutrition disorders) | 86 | 13
Hypoalbuminaemia (Metabolism and nutrition disorders) | 47 | 12
Hypokalaemia (Metabolism and nutrition disorders) | 28 | 6
Hyponatraemia (Metabolism and nutrition disorders) | 25 | 6
Hypophosphataemia (Metabolism and nutrition disorders) | 13 | 4
Back pain (Musculoskeletal and connective tissue disorders) | 29 | 9
Pain in extremity (Musculoskeletal and connective tissue disorders) | 27 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 24 | 6
Headache (Nervous system disorders) | 74 | 7
Dizziness (Nervous system disorders) | 39 | 4
Insomnia (Psychiatric disorders) | 17 | 6
Proteinuria (Renal and urinary disorders) | 114 | 26
Cough (Respiratory, thoracic and mediastinal disorders) | 43 | 10
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 28 | 0
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 144 | 5
Rash (Skin and subcutaneous tissue disorders) | 35 | 6
Hypertension (Vascular disorders) | 123 | 18

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
All clinical study findings and documents will be regarded as confidential. The investigator and members of his/her research team must not disclose such information without prior written approval from the sponsor.

DOCUMENTS (2):
  • Study Protocol (2017-03-10): https://cdn.clinicaltrials.gov/large-docs/60/NCT02329860/Prot_000.pdf
  • Statistical Analysis Plan (2019-07-18): https://cdn.clinicaltrials.gov/large-docs/60/NCT02329860/SAP_001.pdf